CLINICAL TRIAL: NCT05909332
Title: A Randomized, Open-label Phase III Clinical Trial Comparing Antivascular Therapy Combined With Standard Chemotherapy and Standard Chemotherapy in Adjuvant Therapy for Patients With Triple-Negative Breast Cancer, Basal-like Immunosuppressed Subtype (BCTOP-T-A03)
Brief Title: Study of Antivascular Therapy Combined With Chemotherapy Versus Chemotherapy in Adjuvant Therapy of TNBC-BLIS Patients (BCTOP-T-A03)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCTOP-T-A03
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: triple negative breast cancer; adjuvant therapy; antivascular therapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-A (Experimental): BP102 (10 mg/kg) iv D1 and D15 repeated administration of Q4W + Chemotherapy ddEC-P(described below). This was followed by maintenance therapy with BP102 (10 mg/kg) iv D1 and D15 repeated administration of Q4W to complete treatment with a total duration of 1 year from the first dose.
  Chemotherapy: ddEC-P (dose-dense Epirubicin and Cyclophosphamide followed by Nab-paclitaxel). Epirubicin (75-100 mg/m2) iv D1 + Cyclophosphamide (600 mg/m2) iv D1 repeated administration of Q2W for a total of 4 doses, followed by Nab-paclitaxel (125 mg/m2) once weekly (QW) for 4 weeks.
  Interventions: Drug: Antivascular therapy; Drug: Chemotherapy
- Arm-B (Active Comparator): Chemotherapy: ddEC-P (dose-dense Epirubicin and Cyclophosphamide followed by Nab-paclitaxel). Epirubicin (75-100 mg/m2) iv D1 + Cyclophosphamide (600 mg/m2) iv D1 repeated administration of Q2W for a total of 4 doses, followed by Nab-paclitaxel (125 mg/m2) once weekly (QW) for 4 weeks.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Antivascular therapy — BP102 (anti VEGFR)
  Arms: Arm-A
Drug: Chemotherapy — ddEC-P

SUMMARY:
This is a randomized, open-label phase III clinical trial comparing antivascular therapy combined with standard chemotherapy and standard chemotherapy in adjuvant therapy for patients with triple-negative breast cancer, basal-like/Immune suppressed subtype.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70 years old;
* Eastern Oncology Collaborative Group (ECOG) physical status score: 0 or 1;
* Histological results recorded as TNBC (negative HER2, ER, and PgR status) and BLIS subtype according to the classification of FUSCC;
* Have stage IIA-IIIIC triple-negative breast cancer with non-metastatic surgically treated: pT1-3N1-3M0;
* Adequate hematological and end-organ function as defined by the following laboratory test results, which need to be completed within 28 days prior to the first study treatment: absolute neutrophil count (ANC) ≥ 1500 cells/μL (no G-CSF support therapy within 2 weeks prior to day 1 of course 1); Platelet count ≥ 75×109/L (no platelet transfusion within 2 weeks before day 1 of course 1); hemoglobin ≥ 9.0 g/dL (no RBC transfusion within 2 weeks before day 1 of course 1); AST, ALT, and alkaline phosphatase ≤ 3 × upper limit of normal (ULN) serum total bilirubin ≤ 1.0 × ULN; serum creatinine ≤ 1ULN and with an endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula);
* The surgical incision had fully healed prior to the commencement of the study;
* Female participants of reproductive potential are required to use a medically accepted form of contraception during the course of the study treatment and for at least three months following the last administration of the investigational drug;
* Sign the Informed Consent Form (ICF). The patient is judged by the investigator to have the ability to comply with the provisions of the protocol.

Exclusion Criteria:

* Has received neoadjuvant therapy (including chemotherapy, targeted therapy, and radiotherapy)
* Has bilateral breast cancer;
* Has a previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
* Has metastatic (Stage 4) breast cancer;
* Has any >T4 lesion (UICC1987) (with skin involvement, mass adhesion and fixation, and inflammatory breast cancer);
* Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (a cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous to randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
* Is pregnant, breastfeeding women, or women of childbearing age who cannot practice effective contraceptives;
* Patients participating in other clinical trials at the same time;
* Has known allergy to taxane and excipients.
* Has severe or uncontrolled infection;
* Has a history of psychotropic substance abuse and was unable to abandon drug habits or those with a history of mental disorders;
* the researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
iDFS | 5 years
  invasive disease-free survival

SECONDARY OUTCOMES:
DRFS | 5 years
  distant recurrence free survival
OS | 5 years
  overall survival
AE | 5 years
  adverse effects

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Academy of Medical Sciences Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangdong, Guangzhou
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided